CLINICAL TRIAL: NCT00002429
Title: Evaluation of HIV RNA Suppression Produced by a Triple Combination Regimen Containing an Enteric Coated Formulation of Didanosine (ddI EC) Administered Once Daily Compared to a Reference Combination Regimen
Brief Title: Evaluation of an Anti-HIV Drug Combination That Includes a Coated Form of Didanosine (ddI EC) Compared to a Typical Anti-HIV Drug Regimen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 039F; AI454-152
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2011-04

CONDITIONS: HIV Infections
Keywords: Didanosine; Drug Therapy, Combination; Stavudine; RNA, Viral; Nelfinavir; Reverse Transcriptase Inhibitors; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — lamivudine, zidovudine drug combination; Nelfinavir; Stavudine; Didanosine

INTERVENTIONS:
Drug: Lamivudine/Zidovudine
Drug: Nelfinavir mesylate
Drug: Stavudine
Drug: Didanosine

SUMMARY:
This study tests a new form of didanosine, ddI EC, a coated pill that passes through the stomach before dissolving. The purpose of this study is to compare the effectiveness of an anti-HIV drug combination that includes ddI EC versus another anti-HIV drug combination.

DETAILED DESCRIPTION:
Patients are randomized to 1 of 2 groups for 48 weeks of open-label treatment. Group 1 receives ddI EC plus d4T plus NFV. Group 2 receives Combivir plus NFV. Antiviral activity is determined by the proportion of patients with HIV RNA levels of less than 400 copies/ml at Week 48.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have a viral load of at least 2,000 copies/ml and a CD4 count of at least 200 cells/mm3.
* Are at least 18 years old.
* Agree to practice sexual abstinence or to use effective barrier methods of birth control (such as condoms).

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have had severe diarrhea within 30 days of study entry.
* Have a history of pancreatic disease or any other serious condition.
* Have hepatitis within 30 days of study entry.
* Are diagnosed with an opportunistic (AIDS-related) infection at the time of enrollment.
* Are unable to take medications by mouth.
* Have received certain medications.
* Are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 1999-07; Primary Completion 2001-01 (Actual); Study Completion 2001-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (23):
- United States (20):
  - Sorra Research Ctr / Med Forum, Birmingham, Alabama
  - Body Positive, Phoenix, Arizona
  - AIDS Healthcare Foundation, Los Angeles, California
  - San Francisco Gen Hosp, San Francisco, California
  - Med Alternatives, Fort Lauderdale, Florida
  - County Line Med CtrInc, Pembrook, Florida
  - Dr Gerald Pierone Jr, Vero Beach, Florida
  - The CORE Ctr, Chicago, Illinois
  - Indiana Univ Med Ctr, Indianapolis, Indiana
  - Univ of Kansas School of Medicine, Wichita, Kansas
  - Henry Ford Hosp, Detroit, Michigan
  - Dartmouth-Hitchcock Med Ctr, Lebanon, New Hampshire
  - NJCRI, Newark, New Jersey
  - Infectious Disease Assoc of Central Jersey, Somerville, New Jersey
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Anderson Clinical Research, Pittsburgh, Pennsylvania
  - Univ of Texas Southwestern Med Ctr of Dallas, Dallas, Texas
  - Gathe, Joseph, M.D., Houston, Texas
  - Montrose Clinic, Houston, Texas
  - Hampton Roads Med Specialists, Hampton, Virginia
- Canada (3):
  - Clinique Medicale du Quartier Latin, Montreal, Quebec
  - Clinique Medicale L'Actuele, Montreal, Quebec
  - Dr Roger P Leblanc, Montreal, Quebec

REFERENCES:
- [Background] Gathe J, Badero R, Grimwood A, Abrams L, Klesczewski K, Mclaren C. AI454152: Comparison of a Triple Combination Regimen Containing an Enteric Coated Formulation of Didanosine Administered Once-Daily Versus a Regimen of Combivir Plus Nelfinavir. 8th Conference on Retroviruses and Opportunistic Infections, 2001 Feb 4-8. (abstract no 319)